CLINICAL TRIAL: NCT07176975
Title: Phase I Open-label, Dose Escalation and Expansion Trial of BI 1831169 in Combination With an Anti-PD1 mAb in Japanese Patients With Advanced/Metastatic Solid Tumours
Brief Title: A Study to Test How Well Different Doses of BI 1831169 in Combination With an Anti-PD1 Antibody Are Tolerated in Japanese People With Different Advanced Cancers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1456-0004; U1111-1294-3482 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2025-09-15; First posted 2025-09-16 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumors
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Dose escalation part: BI 1831169 dose level 1 + anti-PD-1 antibody (Experimental)
  Interventions: Drug: BI 1831169; Drug: nivolumab
- Dose escalation part: BI 1831169 dose level 2 + anti-PD-1 antibody (Experimental)
  Interventions: Drug: BI 1831169; Drug: nivolumab
- Dose escalation part: BI 1831169 dose level 3 + anti-PD-1 antibody (Experimental)
  Interventions: Drug: BI 1831169; Drug: nivolumab
- Dose escalation part: BI 1831169 dose level 4 + anti-PD-1 antibody (Experimental)
  Interventions: Drug: BI 1831169; Drug: nivolumab
- Dose expansion part: BI 1831169 + anti-PD-1 antibody (Experimental)
  Interventions: Drug: BI 1831169; Drug: nivolumab

INTERVENTIONS:
Drug: BI 1831169 — BI 1831169
Drug: nivolumab — nivolumab

SUMMARY:
This study is open to Japanese adults with different types of advanced cancer (solid tumors). People can join the study if their cancer has spread, and previous treatments were not successful or no treatments exist.

The purpose of this study is to find the highest dose of a medicine called BI 1831169 that people can tolerate when taken together with an anti-PD1 antibody. The anti-PD1 antibody is already used to treat different cancers. Participants receive BI 1831169 together with an anti-PD1 antibody, which is given as an infusion into a vein for up to 1 year.

Participants visit the study site regularly. The number of site visits vary based on the study part and treatment response. Some visits include an overnight stay. The doctors regularly check the participants' health and monitor the tumors. The doctors also take note of any health problems that could have been caused by the study treatment.

ELIGIBILITY:
Inclusion criteria

* Histologically or cytologically confirmed diagnosis of advanced/metastatic solid tumours
* Has at least 1 accessible lesion with a minimum lesion diameter (≥1 cm) for injection of BI 1831169. Lesions must either be easily accessible, or, if not easily accessible, patients must be willing to undergo repeat procedures for injections of BI 1831169.
* Has failed conventional treatment or for whom no therapy of proven efficacy exists or who is not eligible for established treatment options. Patients must have exhausted available treatment options known to prolong survival for their disease.
* Medically fit and willing to undergo all mandatory trial procedures
* Eastern Cooperative Oncology Group (ECOG) Score of 0 or 1, and life expectancy of at least ≥3 months after the start of the treatment, according to the investigator's judgement
* Adequate organ function or bone marrow reserve as demonstrated at screening by the following laboratory values:

  * Absolute neutrophil count ≥1.5x10^9/L (≥1.5x10^3/μL, ≥1500/mm^3) without white blood cell growth factor support within 4 weeks of start of trial treatment; platelet count ≥100·10^9/L (≥100·10^3/μL, ≥100·10^3/mm^3), without platelet transfusion within 2 weeks of start of trial treatment
  * Haemoglobin ≥90 g/L (≥9.0 g/dL, ≥5.6 mmol/L)
  * Creatinine ≤1.5x upper limit of normal (ULN)
  * aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3x ULN if no demonstrable liver metastases, or otherwise ≤5x ULN if transaminase elevation is attributable to liver metastases
  * Total bilirubin ≤1.5x ULN, except for patients with Gilbert's syndrome: total bilirubin ≤3.0x ULN or direct bilirubin ≤1.5x ULN
  * Partial thromboplastin time (PTT)/activated partial thromboplastin time (aPTT) <1.5x ULN unless on a stable dose of an anticoagulant and no unexplained elevation of international normalised ratio (INR)
* All toxicities related to previous anti-cancer therapies (including immune related adverse event (irAEs)) have resolved to Common Terminology Criteria for Adverse Events (CTCAE) Grade ≤1 prior to the start of trial treatment (except for alopecia, xerostomia, and immunotherapy related endocrinopathies which may be included if clinically stable on hormone supplements or antidiabetic drugs as per investigator judgement) and others per investigator judgement.
* Male or female, ≥18 years of age at the time of signature of the informed consent form (ICF) Further inclusion criteria apply.

Exclusion criteria

* Major surgery (major according to the investigator's assessment) performed within 4 weeks prior to start of trial treatment
* Radiotherapy within 4 weeks prior to the start of trial treatment, except in case of a brief course of palliative radiotherapy (e.g. for analgesic purpose or for lytic lesions at risk of fracture) which can then be completed within 2 weeks prior to start of trial treatment. Note: No radiation must have been given to any lesions planned to be injected within 6 months of start of treatment.
* Presence of brain metastases unless patient has completed brain radiotherapy and is asymptomatic. Symptomatic brain metastases, untreated malignant brain tumours and/or carcinomatous meningitis are excluded.
* Presence of other active invasive cancers other than the one to be treated in this trial within 3 years prior to screening, except for appropriately treated basal-cell carcinoma of the skin, in situ carcinoma of the uterine cervix, or other local tumours considered cured by local treatment
* Persistent toxicity from previous treatments (including irAEs) that has not resolved to Grade ≤1, except for alopecia, xerostomia, CTCAE Grade 2 neuropathy, asthenia/fatigue, or Grade 2 endocrinopathies controlled by replacement therapy
* Active or chronic hepatitis B or C infection, e.g. Hepatitis B surface antigen (HBsAg) positive or Hepatitis C antibody (anti-HCV) positive (except if hepatitis C virus (HCV)-ribonucleic acid (RNA) negative)
* Patients with history of human immunodeficiency virus (HIV) infection who meet 1 or more of the following criteria:

  * cluster of differentiation 4 (CD4+) count <350 cells/μL
  * Viral load >400 copies/mL (local lab assessment)
  * Not receiving antiretroviral therapy
  * Receiving established antiretroviral therapy for less than 4 weeks prior to the start of study treatment
  * History of AIDS-defining opportunistic infections within 12 months prior to start of study treatment Patients with a history of HIV who do not meet any of the criteria above are eligible to participate but the patient must be under the care of an HIV/Infectious Diseases specialist or an HIV/Infectious Diseases specialist must be consulted prior to inclusion.
* Any severe or serious, acute or chronic medical or psychiatric condition or laboratory abnormality as per investigator's judgement that may increase the risk associated with trial participation or investigational medicinal product (IMP) administration, including ongoing or active infection requiring systemic antibiotics Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2026-02-12 (Estimated); Primary Completion 2029-01-15 (Estimated); Study Completion 2029-05-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of dose limiting toxicities (DLTs) during the maximum tolerated dose (MTD) evaluation period | up to 6 weeks

SECONDARY OUTCOMES:
Occurrence of dose limiting toxicities (DLTs) during the on-treatment period. | up to 12 months
Occurrence of adverse events (AEs) during the on-treatment period | up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center Hospital East, Chiba, Kashiwa, Japan

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section 'time frame' are fulfilled, researchers can use the following link https:// www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents -upon signing of a 'Document Sharing Agreement'.For study data -1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor'spublication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com